CLINICAL TRIAL: NCT03575702
Title: International, Multicenter, Open-label, Randomized, Comparative Clinical Study of Efficiency and Safety of Medicinal Product Uritos® (Imidafenacin, Film-coated Tablets; 0,1 mg, Kyorin Pharmaceutical Co. Ltd, Japan) and Urotol® (Tolterodine, Film-coated Tablets 2 mg, Zentiva k.s., Czech Republic) for Treatment of Overactive Bladder
Brief Title: Efficacy and Safety Evaluating Study to Compare Uritos® (Imidafenacin) and Urotol® (Tolterodine) for Treatment of Overactive Bladder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Synergy Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG04043028
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; urinary incontinence; frequent urination; urge incontinence; urgency episodes
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urinary Incontinence, Urge | interventions — imidafenacin; Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uritos® (Experimental): one tablet orally twice a day (after breakfast and dinner) for 12 weeks
  Interventions: Drug: Uritos®
- Urotol® (Active Comparator): one tablet orally twice a day (after breakfast and dinner) for 12 weeks
  Interventions: Drug: Urotol®

INTERVENTIONS:
Drug: Uritos® — film-coated tablets 0.1 mg
  Other Names: Imidafenacin
  Arms: Uritos®
Drug: Urotol® — film coated tablets, 2 mg
  Other Names: Tolterodine
  Arms: Urotol®

SUMMARY:
Objective of this study was confirmation on non-inferiority and validation of similar safety profile of new anti-muscarinic medicinal product Uritos® (Imidafenacin) in comparison with other product from m-cholinergic antagonists group Urotol® (Tolterodine).

DETAILED DESCRIPTION:
To assess clinical efficiency and safety of Uritos® (Imidafenacin) in comparison to Urotol® (Tolterodine) according to its influence on urination frequency and number of urinary incontinence episodes a total of 327 patients underwent screening and 300 patients were randomized (150 patients in the Uritos® group and 150 patients in the Urotol® group). Screening period was not exceeding 2 weeks (14 days). Therapy was performed during 12 weeks (84 days). Every patient received only one treatment (Uritos® or Urotol®) during the treatment period. Patients were returning to the trial site to assessment visits on Weeks 2, 4, 8 and 12 with permissible variation ± 3 days. Observation period after the end of treatment - 30 ± 5 days (could be performed through telephone connection without need for physician appointment by patient). Maximum observation period: 136 days.

Efficacy and safety parameters were assessed as per primary and secondary endpoints.

The results of this study could potentially provide new optimum approaches to OAB treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed dated informed consent.
2. Confirmed overactive bladder (OAB). The OAB diagnosis was made based on characteristic symptoms of the patient:

   1. urinary incontinence - 5 or more episodes a week;
   2. frequent urination - 8 or more times a day;
   3. imperative urination urge - 1 or more episodes a day.
3. The duration of the presence of OAB symptoms is 3 months or more (the assessment is based on patient's history and medical records).
4. Overactive bladder Awareness Tool Questionnaire (OAB Awareness Tool) score 8 and more at the screening visit and randomization visit.
5. Negative result of the urine pregnancy test at the screening and the randomization visit before receiving the first dose of the study drug in women of childbearing potential.
6. Female patients of childbearing potential and male patients and their female partners should use at least two birth control methods, one of those is barrier, during the entire study period and for at least 35 days following administration of the last dose of the study product. Acceptable methods of contraception:

   * oral, transdermal, implantation or injection hormone therapy;
   * effective intrauterine devices;
   * double barrier contraceptive methods.
7. Willingness and ability to follow the study visits schedule, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. A history of hypersensitivity or suspected hypersensitivity to tolterodine or imidafenacin.
2. Structural abnormalities of the bladder, including bladder cancer, bladder stones, interstitial cystitis.
3. The volume of residual urine is 100 ml or more with bladder ultrasound.
4. Documented diagnosis of stress urinary incontinence.
5. Operative interventions on the bladder or urethra within the previous 6 months or indications for surgical treatment for OAB.
6. Exacerbation of gynecological diseases including endometriosis, uterine leiomyoma exceeding 3 cm in diameter.
7. Prostate cancer.
8. Prostate diseases with clinically significant urodynamics abnormality (benign prostatic hyperplasia, acute and chronic prostatitis, prostatic calculus).
9. Renal and urinary inflammatory disorders (pyelonephritis, bacterial cystitis, urethritis).
10. For male, the prostatic specific antigen (PSA) level above 4 ng/mL.
11. Severe liver impairment alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) level 3 and more times exceeding the upper limit of normal and/or total bilirubin level 1.5 times exceeding the upper limit of normal.
12. Moderate or severe renal impairment based on the medical records and/or glomerular filtration rate < 50 mL/min determined by Cockroft-Gault formula and/or blood creatinine level > 133 μmol/L at screening.
13. A positive test result for hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
14. Patients suffering from a neoplastic condition without remission at least within 5 years from the start of administration of the study product.
15. Vascular dementia, dementia in Alzheimer's disease, dementia in other diseases, including organic amnestic syndrome.
16. Parkinson's disease or secondary parkinsonism.
17. Nonspecific ulcerative colitis, including severe ulcerative colitis.
18. Thyroid disorders with hyperthyroidism signs.
19. Chronic heart insufficiency Stage III-IV by New York Heart Association Chronic heart insufficiency classification (NYHA).
20. Hypotension: systolic blood pressure (SBP) < 90 mm Hg and/or diastolic blood pressure (DBP) < 60 mm Hg.
21. Uncontrolled medically induced hypertension.
22. Hemodynamically and/or clinically significant heart arrhythmias.
23. QTc prolongation up to 450 ms and more in men and 470 ms and more in women.
24. Open-angle glaucoma.
25. Myasthenia gravis.
26. Megacolon, paralytic ileus, pyloric part of the stomach/duodenal occlusion and any other conditions associated with clinically significant gastric/intestinal obstruction or depressed motility.
27. Necessity of intake and/or intake of prohibited products listed in the Section "Acceptable and prohibited recent and concomitant therapy" within 7 days before the start of therapy.
28. Drug abuse, chronic alcoholism, any psychotic disorders.
29. Participation in other studies within 3 months prior to the beginning of the current study and/or during participation in this study.
30. Pregnancy and/or breastfeeding.
31. Female patients of childbearing potential, having an unprotected sexual contact with a male person non-sterilized by vasectomy during at least 6 months, within 14 days before administration of the study product.
32. Inability to follow protocol procedures.
33. Any other acute or exacerbation and/or decompensation of chronic diseases at inclusion in the study.
34. Patient's behavior, any safety reasons, clinical and administrative reasons, which, according to Investigator's opinion, may potentially affect the study drug safety/efficiency assessment.
35. Other medical and psychiatric conditions or deviations of laboratory parameter which may increase patient risk associated with participation in the study or administration of the study product, or which can influence the interpretation of the study results and, according to Investigator's opinion, make a person ineligible for participation in this study.
36. Patients who are employees of the study site or patients who are employees of the Sponsor/Contract Research Organization (CRO), directly involved in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (11):
- Russia (11):
  - Family polyclinic №4, LLC, Korolyov
  - A.I. Evdokimov Moscow State University of Medicine and Dentistry, Municipal Clinical Hospital named after Spasokukotskiy S.I, Moscow
  - N.I. Pirogov Russian National Research University, Moscow
  - National Medical Radiological Center, Moscow
  - National N.I. Pirogov Medical and Surgical Center, Moscow
  - Rostov State Medical University, Rostov-on-Don
  - All-Russian A.M. Nikiforov Center for Emergency and Radiation Medicine, Saint Petersburg
  - Baltic Medicine LLC, Saint Petersburg
  - I.P. Pavlov First St. Petersburg State Medical University, Saint Petersburg
  - OrKli Hospital, LLC, Saint Petersburg
  - St. Petersburg State-Funded Healthcare Institution St. Luka Clinical Hospital, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrollment was conducted in 11 clinical sites in Russia between July 2016 and April 2017. After the screening period 300 patients (150 in each group) were included in the study. 299 patients started study treatments.
Period: Overall Study
Arm/Group | Uritos® | Urotol®
Started | 149 | 150
Completed | 143 | 146
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Patient non compliance | 4 | 0

BASELINE CHARACTERISTICS:
Population: FAS (Full Analysis Set) population, which included all randomized patients who received at least one dose of the drug and had at least one efficiency evaluation after visit 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Uritos® | Urotol® | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.50) | 46.1 (13.54) | 46.6 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 121 | 245
  Male | 24 | 27 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 146 | 148 | 294
  Asian | 2 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Calculated as patient's weight (kg) / height (m^2)
  kg/m^2 | 25.7 (5.48) | 25.8 (5.33) | 25.8 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Daily Number of Urination Episodes at Week 12
Description: The mean daily number of urination episodes was calculated as the total number of episodes (on the basis of the data that patients entered into their diaries) per day (from 7 am to 7 am the next day) for the study period (between visits) divided by the number of days in the period.
Time Frame: Baseline and Week 12
Population: The efficiency analysis was performed on the FAS (Full Analysis Set) population, which included all randomized patients who received at least one dose of the drug and had at least one efficiency evaluation after visit 2.
Measure: Mean (Standard Deviation); unit: urination episodes per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
urination episodes per day
  Baseline | 12.5 (3.5) | 11.9 (2.7)
  Week 12 of treatment | 9.0 (3.0) | 8.6 (2.5)
  Change | -3.6 (3.0) | -3.4 (2.6)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; The null hypothesis is that effect of Urotol according to the assessment of mean daily urination episodes exceeds effect of Uritos. A sample containing of 222 patients (111 per study group) is considered sufficient to prove the alternative hypothesis at the significance level 0.025% and study power 80%. Given the expected drop out rate during the treatment period, the total number of patients to be randomized is 300 (150 in each group); Test type: Non-Inferiority — The non-inferiority margin is considered as change in mean daily urination episodes of 0,8 episodes per day; p = 0.5595, ANCOVA; The number of urination episodes at the initiation of therapy is used as covariate, and the therapy group is used as a factor; Mean Difference (Final Values) = 0.17, 95% CI 1-sided [upper limit 0.38], Standard Error of Mean 0.34

2. Secondary Outcome: Change in the Mean Daily Number of Incontinence Episodes at Week 12
Description: The mean daily number of incontinence episodes was calculated as the total number of episodes (on the basis of the data that patients entered into their diaries) per day (from 7 am to 7 am the next day) for the study period (between visits) divided by the number of days in the period.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: incontinence episodes per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
incontinence episodes per day
  Baseline | 2.5 (2.4) | 2.4 (2.3)
  Week 12 of treatment | 0.4 (0.9) | 0.5 (1.2)
  Change | -2.1 (2.2) | -1.9 (1.8)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0008, ANCOVA

3. Secondary Outcome: Change in the Mean Daytime Number of Incontinence Episodes at Week 12
Description: The mean daytime number of incontinence episodes was calculated as the total number of episodes from 7 am to 11 pm for the study period (between visits) divided by the number of days in the period.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: daytime incontinence episodes per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
daytime incontinence episodes per day
  Baseline | 2.0 (1.9) | 1.9 (1.8)
  Week 12 of treatment | 0.4 (0.7) | 0.4 (0.9)
  Change | -1.7 (1.7) | -1.5 (1.4)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0099, ANCOVA

4. Secondary Outcome: Change in the Mean Nighttime Number of Incontinence Episodes at Week 12
Description: The mean nighttime number of incontinence episodes was calculated as the total number of episodes from 11 pm to 7 am for the study period (between visits) divided by the number of days in the period.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nighttime incontinence episode per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
nighttime incontinence episode per day
  Baseline | 0.5 (0.8) | 0.5 (0.8)
  Week 12 of treatment | 0.1 (0.3) | 0.1 (0.4)
  Change | -0.4 (0.8) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p < 0.0001, ANCOVA

5. Secondary Outcome: Change in the Mean Number of Incontinence Episodes at Week 2, 4 and 8
Description: Separately for daily, daytime and nighttime measurements.
Time Frame: Baseline and Week 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: incontinence episodes per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
incontinence episodes per day
  Baseline number of daily incontinence episodes | 2.5 (2.4) | 2.4 (2.3)
  Change in daily incontinence episodes (week 2) | -1.5 (1.8) | -1.3 (1.3)
  Change in daily incontinence episodes (week 4) | -1.8 (2.0) | -1.7 (1.5)
  Change in daily incontinence episodes (week 8) | -2.0 (2.0) | -1.8 (1.5)
  Baseline number of daytime incontinence episodes | 2.0 (1.9) | 1.9 (1.8)
  Change in daytime incontinence episodes (week 2) | -1.2 (1.3) | -1.0 (1.1)
  Change in daytime incontinence episodes (week 4) | -1.5 (1.5) | -1.3 (1.3)
  Change in daytime incontinence episodes (week 8) | -1.7 (1.5) | -1.4 (1.3)
  Baseline number of nightime incontinence episodes | 0.5 (0.8) | 0.5 (0.8)
  Change in nighttime incontinence episodes (week 2) | -0.3 (0.6) | -0.3 (0.5)
  Change in nighttime incontinence episodes (week 4) | -0.3 (0.8) | -0.4 (0.6)
  Change in nighttime incontinence episodes (week 8) | -0.3 (0.7) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p < 0.0001, ANCOVA; Changes in number of daily incontinence episodes - week 2
Statistical Analysis 2: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0236, ANCOVA; Changes in number of daily incontinence episodes - week 4
Statistical Analysis 3: Comparison: Uritos® vs Urotol®; Test type: Other; p < 0.0001, ANCOVA; Changes in number of daily incontinence episodes - week 8
Statistical Analysis 4: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0018, ANCOVA; Changes in daytime number of daily incontinence episodes - week 2
Statistical Analysis 5: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.3835, ANCOVA; Changes in daytime number of daily incontinence episodes - week 4
Statistical Analysis 6: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0088, ANCOVA; Changes in daytime number of daily incontinence episodes - week 8
Statistical Analysis 7: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0004, ANCOVA; Changes in nighttime number of daily incontinence episodes - week 2
Statistical Analysis 8: Comparison: Uritos® vs Urotol®; Test type: Other; p < 0.0001, ANCOVA; Changes in nighttime number of daily incontinence episodes - week 4
Statistical Analysis 9: Comparison: Uritos® vs Urotol®; Test type: Other; p < 0.0001, ANCOVA; Changes in nighttime number of daily incontinence episodes - week 8

6. Secondary Outcome: Change in the Mean Weekly Number of Incontinence Episodes at Week 12
Description: The mean weekly number of incontinence episodes was calculated as the total number of episodes per day (from 7 am to 7 am the next day) for the study period (between visits) divided by the number of weeks in the period.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: incontinence episodes per week
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
incontinence episodes per week
  Baseline | 17.2 (16.8) | 16.9 (15.7)
  Week 12 of treatment | 3.0 (6.5) | 3.2 (8.3)
  Change | -14.5 (15.3) | -13.6 (12.4)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.0008, ANCOVA

7. Secondary Outcome: Change in the Mean Daily Number of Urination Episodes at Week 2, 4 and 8 Visit as Compared to the Treatment Initiation Visit
Description: as for outcome 2
Time Frame: Baseline and Week 2, 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: urination episodes per day
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
urination episodes per day
  Baseline | 12.5 (3.5) | 11.9 (2.7)
  Week 2 of treatment | 10.6 (2.9) | 10.3 (2.6)
  Change (week 2) | -1.9 (2.6) | -1.6 (2.1)
  Week 4 of treatment | 9.6 (2.7) | 9.4 (2.6)
  Change (week 4) | -2.8 (2.7) | -2.6 (2.3)
  Week 8 of treatment | 9.4 (2.7) | 8.9 (2.4)
  Change (week 8) | -3.2 (2.9) | -3.1 (2.5)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.1348, ANCOVA; Week 2 changes
Statistical Analysis 2: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.3199, ANCOVA; Week 4 changes
Statistical Analysis 3: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.9537, ANCOVA; Week 8 changes

8. Secondary Outcome: Changes in the Overactive Bladder Symptom Score According to Overactive Bladder (OAB) Awareness Tool Questionnaire at 2, 4, 8 and 12 Week
Description: Overactive bladder (OAB) Awareness Tool Questionnaire (version OAB-V8, containing 8 questions) is a validated questionnaire. Patient is asked to answer 8 questions concerning typical symptoms of OAB giving answers with a scale with minimum - 0 score defined as "no bothering at all" and maximmum - 5 score defined as "a very big deal" to assess the severity of these symptoms. All answers are simply summed to make a combined final score. Male participants should add 2 points to their final score. The final scores range from 0 to 40 (for women) and 42 (for men). The score equal to 8 and more is interpreted as high probability of OAB presence, with the higher scores indicating more bothersome symptoms of OAB.
Time Frame: Baseline and Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
scores on a scale
  Baseline | 24.3 (7.5) | 23.8 (7.1)
  Change (week 2) | -8.0 (8.2) | -8.2 (6.6)
  Change (week 4) | -10.6 (7.7) | -10.8 (6.9)
  Change (week 8) | -12.4 (8.5) | -13.0 (8.0)
  Change (week 12) | -14.2 (8.5) | -14.5 (8.0)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.5321, t-test, 1 sided; Change week 12

9. Secondary Outcome: Change in the EQ-5D-based Quality of Life at Week 12
Description: The Euro Quality of Life five Dimensions questionnaire ( EQ-5D, version EQ-5D-5L) is a validated questionnaire for the assessment of health-related quality of life. It consists of a questionnaire and a visual analogue scale (EQ-VAS). The self-assessment questionnaire is self-reported description of the subject's current health in 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The subject is asked to assess their own current level of function in each dimension by 5-level scale from "no problems" to "significant problem" grades. The EQ-VAS is a self-rated health status using a VAS in mm from 0 (the worse health status) to 100 (the best health status). The EQ-VAS records the subject's perceptions of their own current overall health quantitatively in mm and can be used to monitor changes with time. The results of patients assessment by VAS are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale, mm
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 148 | 148
score on a scale, mm
  Baseline | 67.7 (13.9) | 66.8 (15.0)
  Week 12 of treatment | 81.7 (13.4) | 79.5 (15.4)
  Change (week 12) | 13.8 (15.5) | 12.5 (14.7)
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.4839, t-test, 1 sided; Change week 12

10. Other Pre Specified Outcome: Number of Patients With Adverse Events (AEs)
Time Frame: Up to 35 days after the end of treatment
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Count of Participants; unit: Participants
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
Participants | 70 | 72
Statistical Analysis 1: Comparison: Uritos® vs Urotol®; Test type: Other; p = 0.86, Chi-squared

11. Other Pre Specified Outcome: Number of Patients With Serious Adverse Events (SAEs)
Time Frame: Up to 35 days after the end of treatment
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Count of Participants; unit: Participants
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
Participants | 0 | 0

12. Other Pre Specified Outcome: Changes in the Volume of Residual Urine
Description: Measured via the urine bladder ultrasound (US)
Time Frame: Baseline and Week 4, 8 and 12
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
ml
  Baseline | 10.0 (10.2) | 10.6 (11.3)
  Change week 4 of treatment | -0.9 (10.9) | -1.3 (10.8)
  Change week 8 of treatment | -1.4 (12.7) | -2.2 (12.5)
  Change week 12 of treatment | -1.5 (12.6) | -2.0 (13.0)

13. Other Pre Specified Outcome: Number of Patients With Clinically Significant Changes in Laboratory Parameters
Description: Including blood chemistry, blood count and urinalysis
Time Frame: Week 8 and 12
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Count of Participants; unit: Participants
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
Participants
  Week 8 of treatment | 2 | 1
  Week 12 of treatment | 1 | 3

14. Other Pre Specified Outcome: Number of Patients With Clinically Significant Changes in ECG Parameters
Time Frame: Week 12 of treatment
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Count of Participants; unit: Participants
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
Participants | 0 | 0

15. Other Pre Specified Outcome: Number of Patients With Clinically Significant Vital Signs Changes
Time Frame: Week 12 of treatment
Population: Safety Population - All randomized patients taken at least one dose of investigational/reference drug
Measure: Count of Participants; unit: Participants
Arm/Group | Uritos® | Urotol®
Number analyzed (Participants) | 149 | 150
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 35 days after the end of treatment
Arm/Group | Uritos® | Urotol®
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/150
Other Adverse Events (participants affected / at risk) | 70/149 | 72/150
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uritos® (N=149) | Urotol® (N=150)
Dry mouth (Gastrointestinal disorders) | 40 (56) | 45 (55)
Nausea (Gastrointestinal disorders) | 13 (15) | 17 (21)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (9)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 11 (15) | 17 (18)
Dizziness (Nervous system disorders) | 5 (6) | 8 (10)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 8 (8) | 11 (11)
Asthenia (General disorders) | 1 (1) | 3 (3)
Thirst (General disorders) | 2 (4) | 1 (2)
Malaise (General disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 4 (4) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 4 (6)
Urinary retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Hypertensive crisis (Vascular disorders) | 1 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03575702/Prot_SAP_000.pdf